CLINICAL TRIAL: NCT02129569
Title: Family-Centered Intervention for the Transition to Living With Multiple Myeloma as a Chronic Illness
Brief Title: Psychoeducational and Behavioral Strategies in Reducing Distress and Anxiety in Patients With Multiple Myeloma and Their Family Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE5A13; NCI-2014-00836 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE 5A13 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2017-03-20 (Actual); Status verified 2017-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Behavior Therapy; Counseling; Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (psychoeducational and behavioral interventions) (Experimental): Participants meet with a nurse in-person for approximately 30 minutes to receive information about strategies for cognitive self-management of distress and an individualized walking prescription to gradually increase their walking to 30 minutes per day, 5 times per week. Participants wear a pedometer for at least 3 consecutive days during weeks 1, 6, and 12. Participants are also contacted by the nurse via telephone at 1 and 3 weeks for supplemental counseling support.
  Interventions: Other: Psychoeducational intervention; Behavioral: behavioral intervention; Other: counseling intervention; Other: questionnaire administration; Other: quality-of-life assessment
- Arm II (control) (Active Comparator): Participants meet with a nurse in-person for approximately 20 minutes to receive NCI educational booklets and a link to the ACS website. Participants are also contacted by the nurse via telephone at 1 and 3 weeks but the calls are primarily social in nature and do not include counseling support.
  Interventions: Other: educational intervention; Other: telephone-based intervention; Other: questionnaire administration; Other: quality-of-life assessment

INTERVENTIONS:
Other: Psychoeducational intervention — Receive information about strategies for cognitive self-management of distress
  Arms: Arm I (psychoeducational and behavioral interventions)
Behavioral: behavioral intervention — Receive individualized walking prescription and wear pedometer
  Other Names: Behavior Conditioning Therapy; Behavior Therapy; Behavioral Modification; Behavioral Therapy; Behavioral Treatment
  Arms: Arm I (psychoeducational and behavioral interventions)
Other: counseling intervention — Receive supplemental counseling support over the phone
  Other Names: counseling and communications studies
  Arms: Arm I (psychoeducational and behavioral interventions)
Other: educational intervention — Receive NCI educational booklets and a link to the ACS website
  Other Names: intervention, educational
  Arms: Arm II (control)
Other: telephone-based intervention — Receive calls that are primarily social in nature
  Arms: Arm II (control)
Other: questionnaire administration — Ancillary studies
Other: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies how well psychoeducational and behavioral strategies work in reducing distress and anxiety in patients with multiple myeloma and their family caregivers. Education and walking programs, may be able to reduce distress and anxiety and improve the well-being and quality of life of patients with multiple myeloma and their family caregivers. Understanding how different forms of education and support can promote emotional wellness may help nurse researchers find ways to improve services provided to patients and family members during cancer treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the effect of the intervention, as compared to the control group, on emotional distress, the primary outcome, measured as anxiety in patients with multiple myeloma and their caregivers at the transition.

II. Evaluate the effect, including the effect size, of the intervention, as compared to the control group, on activation for self-management, fatigue, depression, and health-related quality of life (HRQOL) in both patients and caregivers.

III. Assess the feasibility, acceptability, and content integrity of the intervention in patients with multiple myeloma and their family caregivers.

OUTLINE: Participants are randomized to 1 of 2 arms.

ARM I: Participants meet with a nurse in-person for approximately 30 minutes to receive information about strategies for cognitive self-management of distress and an individualized walking prescription to gradually increase their walking to 30 minutes per day, 5 times per week. Participants wear a pedometer for at least 3 consecutive days during weeks 1, 6, and 12. Participants are also contacted by the nurse via telephone at 1 and 3 weeks for supplemental counseling support.

ARM II: Participants meet with a nurse in-person for approximately 20 minutes to receive National Cancer Institute (NCI) educational booklets and a link to the American Cancer Society (ACS) website. Participants are also contacted by the nurse via telephone at 1 and 3 weeks but the calls are primarily social in nature and do not include counseling support.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS: Within 12 months of a new diagnosis of multiple myeloma or less than or equal to 2 cycles of treatment (all stages, with or without treatment)
* PATIENTS: Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to 2
* PATIENTS: Ambulatory with or without an assistive device (cane, walker)
* PATIENTS: Cognitively intact, as evidenced by orientation to person, place, and time
* PATIENTS: Ability to speak, read, and comprehend English
* PATIENTS: Has an identified family caregiver who is willing to participate
* CAREGIVERS: Any family member, who is identified by the patient as his/her caregiver
* CAREGIVERS: ECOG performance status less than or equal to 2
* CAREGIVERS: Ambulatory with or without an assistive device (cane, walker)
* CAREGIVERS: Cognitively intact, as evidenced by orientation to person, place, and time
* CAREGIVERS: Ability to speak, read, and comprehend English
* CAREGIVERS: Has an identified family member who is a patient
* CAREGIVERS: Caregivers do not need to reside with the patient

Exclusion Criteria:

* PATIENTS: Have severe pain (pain score of 7 to 10 on a 0 to 10 scale)
* PATIENTS: Are at high risk for bone fracture or who have a new fracture needing intervention, as determined by the physician
* PATIENTS: Have untreated venous thrombosis, as determined by the physician
* PATIENTS: Have a life expectancy of less than six months, as determined by the physician, and their caregivers
* PATIENTS: Receiving active, concurrent treatment for a prior history of cancer (hormonal therapies allowed)
* CAREGIVERS: Diagnosis of cancer and received cancer treatment within one year
* CAREGIVERS: Medical condition that significantly affects their ability to walk
* PATIENT or CAREGIVER: Is hearing impaired to the degree that they are unable to hear instructions via the phone
* PATIENTS or CAREGIVER: Lives in a skilled nursing facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11-11 (Actual); Primary Completion 2015-04-11 (Actual); Study Completion 2016-08-17 (Actual)

PRIMARY OUTCOMES:
Change in emotional distress in patients measured as anxiety using the Patient-Reported Outcomes Measurement Information System (PROMIS) | Baseline to up to 12 weeks
  A linear mixed model will be used and the model parameters will be estimated by the method of restricted maximum likelihood.

SECONDARY OUTCOMES:
Change in activation for self-management in patients using the Patient Activation Measure (PAM) | Baseline to up to 12 weeks
  A linear mixed model will be used. If there are large numbers of missing values, the parameters will be estimated by utilizing the "pattern mixture model." Should the change be non-linear, the model may be extended to allow for non-linearity. In the case of parametric model assumption violation, the generalized estimating equation approach may be used.
Change in activation for self-management in caregivers using the PAM | Baseline to up to 12 weeks
  A linear mixed model will be used. If there are large numbers of missing values, the parameters will be estimated by utilizing the "pattern mixture model." Should the change be non-linear, the model may be extended to allow for non-linearity. In the case of parametric model assumption violation, the generalized estimating equation approach may be used.
Change in fatigue in patients using the PROMIS | Baseline to up to 12 weeks
  A linear mixed model will be used. If there are large numbers of missing values, the parameters will be estimated by utilizing the "pattern mixture model." Should the change be non-linear, the model may be extended to allow for non-linearity. In the case of parametric model assumption violation, the generalized estimating equation approach may be used.
Change in fatigue in caregivers using the PROMIS | Baseline to up to 12 weeks
  A linear mixed model will be used. If there are large numbers of missing values, the parameters will be estimated by utilizing the "pattern mixture model." Should the change be non-linear, the model may be extended to allow for non-linearity. In the case of parametric model assumption violation, the generalized estimating equation approach may be used.
Change in depression in patients using the PROMIS | Baseline to up to 12 weeks
  A linear mixed model will be used. If there are large numbers of missing values, the parameters will be estimated by utilizing the "pattern mixture model." Should the change be non-linear, the model may be extended to allow for non-linearity. In the case of parametric model assumption violation, the generalized estimating equation approach may be used.
Change in depression in caregivers using the PROMIS | Baseline to up to 12 weeks
  A linear mixed model will be used. If there are large numbers of missing values, the parameters will be estimated by utilizing the "pattern mixture model." Should the change be non-linear, the model may be extended to allow for non-linearity. In the case of parametric model assumption violation, the generalized estimating equation approach may be used.
Change in HRQOL in patients using the PROMIS short form, Global Health | Baseline to up to 12 weeks
  A linear mixed model will be used. If there are large numbers of missing values, the parameters will be estimated by utilizing the "pattern mixture model." Should the change be non-linear, the model may be extended to allow for non-linearity. In the case of parametric model assumption violation, the generalized estimating equation approach may be used.
Change in HRQOL in caregivers using the PROMIS short form, Global Health | Baseline to up to 12 weeks
  A linear mixed model will be used. If there are large numbers of missing values, the parameters will be estimated by utilizing the "pattern mixture model." Should the change be non-linear, the model may be extended to allow for non-linearity. In the case of parametric model assumption violation, the generalized estimating equation approach may be used.
Feasibility of the intervention, assessed via attrition rates | Up to 12 weeks
Acceptability of the intervention, assessed via consent rates | Up to 12 weeks
Satisfaction with the intervention assessed using an exit interview survey | At 12 weeks
Integrity of the intervention, assessed through fidelity monitoring | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan Mazanec, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Comprehensive Cancer Center, Cleveland, Ohio, United States